CLINICAL TRIAL: NCT06554834
Title: Effects of Three Therapeutic Sessions of the Fourth Ventricle Compression Technique and Rib Raising Osteopathic Technique on Autonomic Nervous System Activity Measured by Heart Rate Variability in 109 Healthy Individuals
Brief Title: Effects of Osteopathic Technique on Autonomic Nervous System Activity
Acronym: Osteo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SomaticMed (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOMATIC2024-001
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Dysautonomia
Keywords: Autonomic Nervous System; Osteopathic Medicine; Heart Rate Variability
MeSH Terms: conditions — Autonomic Nervous System Diseases | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: n this study, 109 healthy subjects will be randomly assigned to one of three groups. The first experimental group will receive three 30-minute sessions of osteopathic therapy using both CV4 and RR techniques. The second group will undergo three 30-minute sessions of the CV4 technique alone. The placebo group will undergo a sham procedure using an ultrasound transducer. To assess the impact of these interventions on autonomic nervous system (ANS) function, Heart Rate Variability (HRV) will be measured using specialized equipment in a seated position over a 5-minute duration.
Who Masked: Participant
Masking Description: This study will employ a single-blind design, where participants will be unaware of the specific intervention they receive. However, the investigators and care providers will be informed about the group assignments to ensure proper administration of the interventions. Blinding will be maintained throughout the study to prevent participant bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CV4 + RR Group (Experimental): Participants will undergo three 30-minute sessions of osteopathic therapy combining the Fourth Ventricle Compression (CV4) and Rib Raising (RR) techniques.
  Interventions: Procedure: CV4 + RR; Device: EEG/HRV/RSA (Electroencephalography, Heart Rate Variability, Respiratory Sinus Arrhythmia) Monitoring using Infiniti System
- CV4 Group (Experimental): Participants will receive three 30-minute sessions of osteopathic therapy focusing solely on the Fourth Ventricle Compression (CV4) technique.
  Interventions: Procedure: CV4; Device: EEG/HRV/RSA (Electroencephalography, Heart Rate Variability, Respiratory Sinus Arrhythmia) Monitoring using Infiniti System
- Placebo Group (Placebo Comparator): Participants will undergo a sham procedure involving an ultrasound transducer for three 30-minute sessions, with no therapeutic intervention.
  Interventions: Device: sham ultrasound transducer; Device: Ultrasound Transducer Sham Procedure; Device: EEG/HRV/RSA (Electroencephalography, Heart Rate Variability, Respiratory Sinus Arrhythmia) Monitoring using Infiniti System

INTERVENTIONS:
Procedure: CV4 + RR — Participants in this group will undergo three 30-minute sessions of osteopathic therapy. The intervention will involve a combination of the Fourth Ventricle Compression (CV4) technique and the Rib Raising (RR) technique. These sessions will be administered once per week over three consecutive weeks. The CV4 technique involves gentle compression of the occiput to influence cranial rhythmic impulses, while the RR technique involves mobilization of the rib cage to impact autonomic nervous system function.
  Arms: CV4 + RR Group
Procedure: CV4 — Participants in this group will receive three 30-minute sessions focusing solely on the Fourth Ventricle Compression (CV4) technique. The sessions will be conducted once per week for three consecutive weeks. The CV4 technique involves applying gentle pressure to the occiput with the goal of affecting cranial rhythmic impulses and promoting autonomic nervous system balance.
  Arms: CV4 Group
Device: sham ultrasound transducer — Participants in the placebo group will undergo three 30-minute sessions of a sham procedure using an ultrasound transducer. The transducer will be applied in a manner that mimics a therapeutic intervention, but without delivering any actual therapeutic effect. These sessions will also be conducted once per week for three consecutive weeks.
  Arms: Placebo Group
Device: Ultrasound Transducer Sham Procedure — Participants in the placebo group will undergo three 30-minute sessions using an ultrasound transducer as part of a sham procedure. The transducer will be applied to the body in a manner that mimics a therapeutic intervention, but it will not deliver any actual therapeutic effect. This procedure is designed to simulate the experience of receiving treatment without providing the physiological benefits associated with active ultrasound therapy. The sessions will be conducted once per week over three consecutive weeks.
  Arms: Placebo Group
Device: EEG/HRV/RSA (Electroencephalography, Heart Rate Variability, Respiratory Sinus Arrhythmia) Monitoring using Infiniti System — Participants in this study will undergo monitoring of Heart Rate Variability (HRV), and Respiratory Sinus Arrhythmia (RSA) using the Infiniti 8 measuring device. This system includes a ProComp Infiniti encoder, which is a versatile and advanced tool for capturing physiological signals, and the Biograph Infiniti software, which, along with the Physiology Suit, allows for detailed analysis and monitoring of autonomic nervous system function.
  Other Names: EEG/HRV/RSA (Electroencephalography, Respiratory Sinus Arrhythmia) Infiniti 8 measuring device, a ProComp Infiniti encoder, and Biograph Infiniti and Physiology Suit software

SUMMARY:
Cranial osteopathic manipulation technique for brain and cranial nerve function, known as the fourth ventricle compression (CV4), has been recognized. Rib raising (RR), aimed at reducing rib restriction and conditions associated with sympathetic hypertonia, is also employed. This study aimed to assess, in about 109 healthy individuals, the effects of osteopathic techniques (CV4 and RR) on autonomic nervous system (ANS) activity, as measured by heart rate variability (HRV).

DETAILED DESCRIPTION:
In this planned study, 109 healthy subjects will be randomly assigned to one of three groups. A total of 90-100 participants are expected to complete all stages of the study, and their data will be used in the final analysis. The first experimental group will undergo three 30-minute sessions of osteopathic therapy, including the CV4 and RR techniques. The second group will receive three 30-minute sessions of the CV4 technique alone. The placebo group will undergo a sham procedure using an ultrasound transducer. To evaluate the impact of these osteopathic techniques on autonomic nervous system (ANS) function, Heart Rate Variability (HRV) will be measured using an EEG/HRV/RSA Infiniti 8 device, ProComp Infiniti encoder, and Biograph Infiniti and Physiology Suit software. Measurements will be conducted in a seated position over a 5-minute duration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years.
* Subjects not currently undergoing any form of rehabilitation, physiotherapy, or osteopathy

Exclusion Criteria:

* Unstable arrhythmia in the patient's history and symptoms related to chest organs (retrosternal pain, difficulty breathing).
* Pregnancy.
* Menstruation.
* Smoking.
* Symptoms suggestive of disorders related to bowel obstruction (bloating with pain, vomiting, diarrhea).
* Surgical treatment in the head.
* Neurological diseases.
* Back and peripheral joint pain, trauma, and musculoskeletal dysfunction in the last 12 months.
* Having undergone physiotherapy or osteopathy treatment within the last month, regardless of the reason

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | Measurements will be taken at three time points: before the intervention (baseline), immediately after the third session (post-intervention), and one month after the final session (follow-up).
  Changes in Heart Rate Variability will be assessed to evaluate the overall autonomic nervous system (ANS) function. HRV will be measured using the standard deviation of normal-to-normal intervals (SDNN) and other relevant time-domain and frequency-domain parameters. Measurements will be taken before the intervention, immediately after the third session, and one month after the final session to evaluate both immediate and sustained effects.
High-Frequency Power (HF) | Measurements will be taken at three time points: before the intervention (baseline), immediately after the third session (post-intervention), and one month after the final session (follow-up).
  The HF component of HRV, which reflects parasympathetic (vagal) activity, will be measured. Changes in HF power will indicate the impact of the osteopathic techniques on parasympathetic regulation. HF power will be expressed in absolute units (ms²) and as a normalized unit.
Low-Frequency Power (LF | Measurements will be taken at three time points: before the intervention (baseline), immediately after the third session (post-intervention), and one month after the final session (follow-up).
  The LF component of HRV, associated with both sympathetic and parasympathetic activity, will be assessed. LF power will be measured to understand its modulation through the interventions. LF power will be reported in absolute units (ms²) and as a normalized unit.
LF/HF Ratio | Measurements will be taken at three time points: before the intervention (baseline), immediately after the third session (post-intervention), and one month after the final session (follow-up).
  The ratio of LF to HF power (LF/HF) will be analyzed as an indicator of the balance between sympathetic and parasympathetic nervous system activity. This measure will help determine the relative predominance of each branch of the autonomic nervous system in response to the osteopathic interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- SomaticMed, Wołomin, Prądzyńskiego, Poland

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns regarding the protection of participant privacy and legal restrictions related to the processing of personal data.